CLINICAL TRIAL: NCT00026117
Title: Phase III Evaluation Of Benefin Shark Cartilage In Patients With Advanced Cancer
Brief Title: Shark Cartilage in Treating Patients With Advanced Colorectal or Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCCTG-971151; CDR0000068987 (Registry Identifier: PDQ (Physician Data Query)); NCCAM
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Colorectal Cancer
Keywords: stage IV colon cancer; stage IV breast cancer; recurrent breast cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Breast Neoplasms, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BeneFin (Experimental): Patients receive oral shark cartilage (BeneFin™) 3-4 times daily. Treatment continues in the absence of unacceptable toxicity. Quality of life is assessed weekly for 1 month and then monthly thereafter during treatment.
  Patients are followed every 6 months for 5 years.
  Interventions: Drug: BenFin
- placebo (Other): Patients receive oral placebo 3-4 times daily. Treatment continues in the absence of unacceptable toxicity. Quality of life is assessed weekly for 1 month and then monthly thereafter during treatment.
  Patients are followed every 6 months for 5 years.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: BenFin
  Arms: BeneFin
Other: placebo
  Arms: placebo

SUMMARY:
RATIONALE: Shark cartilage extract may help shrink or slow the growth of colorectal cancer or breast cancer cells.

PURPOSE: Randomized phase III trial to determine the effectiveness of shark cartilage in treating patients who have advanced colorectal cancer or advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the addition of powdered shark cartilage (BeneFin™) to standard therapy improves overall survival in patients with advanced colorectal or breast cancer.
* Determine whether this therapy has any impact on toxicity in these patients.
* Determine whether this therapy improves the quality of life in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to disease type (breast vs colorectal female vs colorectal male), age (49 and under vs 50-69 vs 70 and over), ECOG performance status (0-1 vs 2), baseline quality of life (UNISCALE rating less than 50% vs 50-75% vs more than 75%), and concurrent chemotherapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Breast or colorectal primary tumor sites

  * Considered incurable
* Breast cancer patients must have disease progression after at least 2 different chemotherapy regimens (may include chemotherapy given as an adjuvant treatment)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Male or female

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hepatic:

* Bilirubin no greater than 3 times upper limit of normal (ULN)

Renal:

* Calcium less than 1.2 times ULN

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Chemotherapy:

* Concurrent chemotherapy allowed
* No concurrent participation in a cytotoxic chemotherapy clinical trial

Other:

* At least 60 days since prior shark cartilage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2001-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 5 years

SECONDARY OUTCOMES:
quality of life | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Loprinzi, MD, Study Chair — Mayo Clinic
Locations (16):
- United States (16):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Duluth, Duluth, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Loprinzi CL, Levitt R, Barton DL, Sloan JA, Atherton PJ, Smith DJ, Dakhil SR, Moore DF Jr, Krook JE, Rowland KM Jr, Mazurczak MA, Berg AR, Kim GP; North Central Cancer Treatment Group. Evaluation of shark cartilage in patients with advanced cancer: a North Central Cancer Treatment Group trial. Cancer. 2005 Jul 1;104(1):176-82. doi: 10.1002/cncr.21107. PMID 15912493